CLINICAL TRIAL: NCT01403818
Title: Pharmacokinetic Study of ASP1941 -A Pharmacokinetic Study to Assess Drug-Drug Interaction Between ASP1941 and Mitiglinide Calcium Hydrate
Brief Title: A Study to Assess the Effect of ASP1941 and Mitiglinide on Their Plasma Concentration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 1941-CL-0074
Record Dates: First submitted 2011-07-25; First posted 2011-07-27 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Healthy; Pharmacokinetics of ASP1941; Pharmacokinetics of Mitiglinide
Keywords: ASP1941; ipragliflozin; Mitiglinide calcium hydrate; Drug-Drug interaction; Pharmacokinetics
MeSH Terms: interventions — ipragliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1 (Experimental): Subjects will receive "ASP1941 alone" and "ASP1941 + Mitiglinide calcium hydrate" in different orders.
  Interventions: Drug: ASP1941; Drug: Mitiglinide calcium hydrate
- Part 2 (Experimental): Subjects will receive "Mitiglinide calcium hydrate alone" and "ASP1941 + Mitiglinide calcium hydrate" in different orders.
  Interventions: Drug: ASP1941; Drug: Mitiglinide calcium hydrate

INTERVENTIONS:
Drug: ASP1941 — oral
  Other Names: ipragliflozin
Drug: Mitiglinide calcium hydrate — oral
  Other Names: Glufast

SUMMARY:
This study is to assess the pharmacokinetic interaction between ASP1941 and Mitiglinide calcium hydrate in healthy volunteers.

DETAILED DESCRIPTION:
This will be a randomized, open label, four group, two-way crossover design study to assess the effect of drug interaction between ASP1941 and Mitiglinide calcium hydrate on the pharmacokinetics of them after separate and concomitant administration to healthy non-elderly adult male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as judged by the investigator/subinvestigator based on the results of physical examinations and laboratory tests
* Body weight ; ≥50.0 kg, <80.0 kg
* Body Mass Index ; ≥17.6, <26.4 kg/m2
* Written informed consent has been obtained

Exclusion Criteria:

* Received any investigational drugs within 120 days before the screening assessment
* Donated 400 mL of whole blood within 90 days, 200 mL of whole blood within 30 days, or d components within 14 days before the screening assessment
* Received medication within 7 days before hospital admission
* A deviation from the assessment criteria of physical examinations or laboratory tests at screening or upon admission
* History of drug allergies
* With renal, hepatic, gastrointestinal, heart, cerebrovascular or respiratory diseases
* Previous treatment with ASP1941

Ages: 20 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of ASP1941 and Mitiglinide calcium hydrate assessed by its plasma concentration change | For up to 72 hours after each administration

SECONDARY OUTCOMES:
Safety assessed by incidence of adverse event, vital signs, 12-lead ECG and laboratory tests | For up to 10 days
Pharmacokinetics of the metabolites of ASP1941 assessed by its plasma concentration change | For 72 hours after ASP1941 administration

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (1):
- Kantou, Japan